CLINICAL TRIAL: NCT05042596
Title: Short Term Outcomes of Fracture Odontoid Management in Assuit University Hospital
Brief Title: Short Term Outcomes of Fracture Odontoid Management
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Shaif Al-Huthaifi, Doctor, Assiut University
Other Study IDs: Outcome of Odontoid fracture
Record Dates: First submitted 2021-09-05; First posted 2021-09-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Spine Injury
Keywords: Odontoid fracture, upper cervical fracture, anterior odontoid screw, NDI.
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate and assess the short-term outcomes of odontoid fracture cases admitted to trauma unit of Assiut university hospital.

DETAILED DESCRIPTION:
patients with completed records, CTs, and Plain radiographs. Sufficient clinical records with documented NDI, The patient will be evaluated in 2 weeks, 6 weeks , and 3 , 6 months post operative .

ELIGIBILITY:
Inclusion Criteria:

* all patients with odontoid fractures admitted to Assiut University Hospital - Department of Orthopedics and Trauma between October 2021 and June 2023

Exclusion Criteria:

* patients who are not available for 6 months follow-up and those with insufficient documentation or records

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient with fracture Odontoid .
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Assess the short term outcomes of Odontoid fracture in skeletally mature patients | 6 months
  To use the NDI as assessment tool of outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad El-Sharkawi, Study Chair — Assiut University; Ahmed Abdelgawaad, Study Director — Assiut University; Mahmoud Ibrahim, Study Director — Assiut University; Ahmed Al-huthaifi, Principal Investigator — Assiut University
Locations (1):
- Assiut UNIVERSITY HOSPITAL, Asyut, Egypt

REFERENCES:
- [Result] Pal D, Sell P, Grevitt M. Type II odontoid fractures in the elderly: an evidence-based narrative review of management. Eur Spine J. 2011 Feb;20(2):195-204. doi: 10.1007/s00586-010-1507-6. Epub 2010 Sep 12. PMID 20835875
- [Result] Wang J, Zheng W, Zhang Z, Li C, Zhou Y. [Percutaneous anterior odontoid and transarticular screw fixation for type II odontoid fractures in elderly patients]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2013 Sep;27(9):1090-3. Chinese. PMID 24279021